CLINICAL TRIAL: NCT00272350
Title: A Phase I/II Trial of ZD6474 for Patients With Recurrent High-Grade and Progressive Low-Grade Gliomas
Brief Title: ZD6474 to Treat Advanced Brain Cancer in Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060063; 06-C-0063; NCT00293566 (obsolete NCT alias)
Record Dates: First submitted 2006-01-05; First posted 2006-01-05 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2014-02-27

CONDITIONS: Recurrent High-Grade Gliomas; Progressive Low-Grade Gliomas; Malignant Gliomas
Keywords: Brain; Tumor; Therapy; Progression; Antiangiogenesis; Brain Tumor; Malignant Glioma
MeSH Terms: conditions — Glioma; Neoplasms; Disease Progression; Brain Neoplasms | interventions — Steroids; vandetanib

INTERVENTIONS:
Drug: Steroids
Drug: ZD6474

SUMMARY:
Background:

In vivo experiments have documented the ability of ZD6474 to inhibit tumor growth in various preclinical tumor models. Given the pronounced neovasculature associated with malignant gliomas, and abundant published data demonstrating the dependence of glioma growth on the maintenance and proliferation of this neovasculature, ZD6474 represents a potentially promising new therapeutic approach to these otherwise refractory tumors.

Thus, we now propose a phase I trial of ZD6474 in patients with recurrent and progressive low-grade gliomas who are on P450-inducing anti-epileptic drugs and a phase II trial for patients with recurrent gliomas not taking P450-inducing anti-epileptic drugs.

Objective:

Phase I - To establish the maximally tolerated dose of ZD6474 and to obtain preliminary information regarding the spectrum of toxicities of ZD6474, and to obtain pharmacokinetic data to patients taking EIAED.

Phase I - To obtain preliminary information regarding potential anti-tumor activity of ZD6474 in patients taking EIAED.

Phase II - To establish data regarding the anti-tumor activity of ZD6474 and to collect information regarding the spectrum of toxicities in patients not taking EIAEDs.

Eligibility:

Patients with histologically proven malignant primary gliomas will be eligible for this protocol. Additionally, patients with progressive low-grade gliomas and patients with infiltrative brain stem gliomas, diagnosed radiographically rather than by biopsy will also be eligible.

Design:

Phase I - Group B patients will be accrued to the formal dose-escalation phase I trial. Groups of patients with recurrent high-grade gliomas will be accrued to increasingly higher doses of ZD6474 until the MTD is established.

Phase II - Patients will be treated at a dose of 300 mg day, every day, on a 4-week cycle.

DETAILED DESCRIPTION:
Background:

In vivo experiments have documented the ability of ZD6474 to inhibit tumor growth in various preclinical tumor models. Given the pronounced neovasculature associated with malignant gliomas, and abundant published data demonstrating the dependence of glioma growth on the maintenance and proliferation of this neovasculature, ZD6474 represents a potentially promising new therapeutic approach to these otherwise refractory tumors.

Thus, we now propose a phase I trial of ZD6474 in patients with recurrent and progressive low-grade gliomas who are on P450-inducing anti-epileptic drugs and a phase II trial for patients with recurrent gliomas not taking P450-inducing anti-epileptic drugs.

Objective:

Phase I - To establish the maximally tolerated dose of ZD6474 and to obtain preliminary information regarding the spectrum of toxicities of ZD6474, and to obtain pharmacokinetic data to patients taking EIAED.

Phase I - To obtain preliminary information regarding potential anti-tumor activity of ZD6474 in patients taking EIAED.

Phase II - To establish data regarding the anti-tumor activity of ZD6474 and to collect information regarding the spectrum of toxicities in patients not taking EIAEDs.

Eligibility:

Patients with histologically proven malignant primary gliomas will be eligible for this protocol. Additionally, patients with progressive low-grade gliomas and patients with infiltrative brain stem gliomas, diagnosed radiographically rather than by biopsy will also be eligible.

Design:

Phase I - Group B patients will be accrued to the formal dose-escalation phase I trial. Groups of patients with recurrent high-grade gliomas will be accrued to increasingly higher doses of ZD6474 until the MTD is established.

Phase II - Patients will be treated at a dose of 300 mg day, every day, on a 4-week cycle.

ELIGIBILITY:
* ELIGIBILITY CRITERIA :

INCLUSION CRITERIA PHASE I:

Patients with histologically proven malignant primary gliomas will be eligible for this protocol. These include glioblastoma multiforme (GBM), gliosarcoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), and malignant glioma/astrocytoma NOS. Additionally, patients with progressive low-grade gliomas and patients with infiltrative brain stem gliomas, diagnosed radiographically rather than by biopsy.

Patients must have an MRI scan performed within 14 days prior to registration.

Patients having undergone recent resection of a recurrent or progressive tumor, will be eligible four weeks after surgery.

Patients must have failed prior radiation therapy.

All patients or their PREVIOUSLY DESIGNATED DPA (if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired is such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study.

Patients must be greater than or equal to 18 years old, and must have a life expectancy greater than 8 weeks.

Patients must have a Karnofsky performance status of greater than or equal to 60.

Patients must be at least six weeks from radiation therapy. Additionally, patients must be at least 6 weeks from nitrosoureas, 4 weeks from temozolomide or carboplatin, 3 weeks from procarbazine, and 2 weeks from last vincristine administration. Patients must be at least 4 weeks from other cytotoxic therapies not listed above and 2 weeks for non-cytotoxic agents (e.g., interferon, tamoxifen) including investigative agents.

Patients must have adequate bone marrow function (WBC greater than or equal to 3,000/microliter ANC greater than or equal to 1,500/mm(3), platelet count of greater than or equal to 100,000/mm(3), and hemoglobin greater than or equal to 10 gm/dl), adequate liver function (SGOT and bilirubin less than or equal to 2 times ULN), and adequate renal function (creatinine less than or equal to 1.5 mg/dL and/or creatinine clearance greater than or equal to 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.

Patients must either not be receiving steroids, or be on a stable dose of steroids for at least five days prior to registration.

Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in remission and off of all therapy for that disease for a minimum of 1 year are ineligible.

This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.

Patients must not be pregnant or nursing, and all patients (both men and women) must be willing to practice birth control during and for 2 months after treatment with ZD6474. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).

A 12 lead electrocardiogram (ECG) to be performed within 2 weeks of trial entry with QTc less than 460 msec.

Only patients on EIAEDs are to be included in Phase I.

A normal echocardiogram to be performed within 2 weeks of trial entry.

EXCLUSION CRITERIA PHASE I:

Any of the following is regarded as a criterion for exclusion from the study:

Patients who, in the view of the treating physician, have significant active hepatic, renal, or psychiatric diseases are ineligible.

Active cardiac disease as defined by:

* Significant cardiac event (including symptomatic heart failure or evidence of cardiac ischemia within 3 months of first dose or presence of any cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
* Clinically significant arrhythmia (multifocal premature ventricular contraction [PVC], bigeminy, trigeminy, ventricular tachycardia, bradycardia) that is symptomatic or requires treatment (CTCAE v3.0 grade 3), or asymptomatic sustained ventricular tachycardia, at the discretion of the investigator.
* Any concurrent medication that may cause QTc prolongation or induce Torsades de Pointes (See Appendix C, Table 1). Drugs listed in Appendix C, Table 2, that in the investigator s opinion cannot be discontinued are allowed; however, must be monitored closely with additional ECGs and laboratory assessments of electrolytes to ensure the patient s safety.
* Previous history of QTc prolongation with other medication.
* Congenital long QT syndrome.
* QTc with Bazett's correction that is unmeasurable, or greater than or equal to 460 msec on screening ECG. If a patient has QTc greater than or equal to 460 msec on screening ECG, a second screen ECG may be repeated at least 24 hours apart. The average QTc from the 2 screening ECGs must be less than 460 msec in order for the patient to be eligible for the study. If the patient meets eligibility requirements in this way, the "baseline" QTc for this patient will be the average of the 3 ECGs (screen 1, screen 2, and pre-1st dose).
* Previous history of left ventricular ejection fraction (LVEF) less than 45 percent as measured by multi-gated acquisition scan (MUGA) or by echocardiogram (ECHO) for patients with previous anthracycline therapy (total dose greater than 450 mg/m(2)) or significant cardiovascular disease or chest irradiation, as determined by the investigator.
* A cardiac arrhythmia serious enough to require therapy (i.e. drugs, AID), angina, symptomatic congestive heart failure and/or a cardiac ejection fraction less than 45 percent.

Prior serious cardiac disease defined as prior coronary bypass surgery, angioplasty, or prior myocardial infarction unless a recent cardiac evaluation (within the last 3 months) demonstrated no significant coronary artery disease (i.e. a negative stress test) and no myocardial wall dysfunction.

Concurrent use of other standard chemotherapeutics or investigative agents or vasoconstrictors for the treatment of migraine (ergotamine, zolmitriptan, sumatriptan) because of the potential for exacerbation of coronary vasoconstriction.

Laboratory results sustained at:

Neutrophils less than 1.5 10(9)/L or platelets less than 100,000/mm(3). Serum creatinine greater than 1.5 x ULRR. Potassium, calcium (ionized calcium or adjusted for albumin), or magnesium concentrations outside normal limits. Supplementation of electrolytes is permitted. Aspartate aminotransferase (AST/SGOT) greater than 2 times ULRR, or AST greater than 5.0 ULRR if judged by the investigator to be related to liver metastases.

Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.

Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg).

Any currently active gastrointestinal disease with diarrhea that may affect the ability of the patient to absorb the ZD6474 or tolerate diarrhea.

Currently pregnant or breast feeding.

Participation in a clinical trial of any investigational agents within 14 days prior to commencing study treatment.

Patients must be at least six weeks from radiation therapy. Additionally, patients must be at least 6 weeks from nitrosoureas, 4 weeks from temozolomide or carboplatin, 3 weeks from procarbazine, and 2 weeks from last vincristine administration. Patients must be at least 4 weeks from other cytotoxic therapies not listed above and 2 weeks for non-cytotoxic agents (e.g., interferon, tamoxifen) including investigative agents.

Any unresolved toxicity greater than CTC (Version 3.0) grade 1 from previous anti-cancer therapy.

INCLUSION CRITERIA PHASE II:

Patients with histologically proven malignant primary gliomas will be eligible for this protocol. These include glioblastoma multiforme (GBM), gliosarcoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), and malignant glioma/astrocytoma NOS.

Patients must have an MRI scan performed within 14 days prior to registration.

Patients having undergone recent resection of a recurrent or progressive tumor, will be eligible four weeks after surgery.

Patients with high-grade gliomas must have failed prior radiation therapy.

All patients or their PREVIOUSLY DESIGNATED DPA (if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study.

Patients must be greater than or equal to 18 years old, and must have a life expectancy greater than 8 weeks.

Patients must have a Karnofsky performance status of greater than or equal to 60.

Patients must be at least six weeks from radiation therapy. Additionally, patients must be at least 6 weeks from nitrosoureas, 4 weeks from temozolomide or carboplatin, 3 weeks from procarbazine, and 2 weeks from last vincristine administration. Patients must be at least 4 weeks from other cytotoxic therapies not listed above and 2 weeks for non-cytotoxic agents (e.g., interferon, tamoxifen) including investigative agents.

Patients must have adequate bone marrow function (WBC greater than or equal to 3,000/microl, ANC greater than or equal to 1,500/mm(3), platelet count of greater than or equal to 100,000/mm(3), and hemoglobin greater than or equal to 10 gm/dl), adequate liver function (SGOT and bilirubin less than or equal to 2 times ULN), and adequate renal function (creatinine less than or equal to 1.5 mg/dL and/or creatinine clearance greater than or equal to 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.

Patients must either not be receiving steroids, or be on a stable dose of steroids for at least five days prior to registration.

Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in remission and off of all therapy for that disease for a minimum of 1 year are ineligible.

This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.

Patients must not be pregnant or nursing, and all patients (both men and women) must be willing to practice birth control during and for 2 months after treatment with ZD6474. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).

A 12 lead electrocardiogram (ECG) to be performed within 2 weeks of trial entry with QTc less than 460 msec.

Only patients taking NEIAEDs are to be included in Phase II.

A normal echocardiogram to be performed within 2 weeks of trial entry.

EXCLUSION CRITERIA PHASE II:

Any of the following is regarded as a criterion for exclusion from the study:

Patients who, in the view of the treating physician, have significant active hepatic, renal, or psychiatric diseases are ineligible.

Active cardiac disease as defined by:

* Significant cardiac event (including symptomatic heart failure or evidence of cardiac ischemia within 3 months of first dose or presence of any cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
* Clinically significant arrhythmia (multifocal premature ventricular contraction [PVC], bigeminy, trigeminy, ventricular tachycardia, bradycardia) that is symptomatic or requires treatment (CTCAE grade 3), or asymptomatic sustained ventricular tachycardia.
* Any concurrent medication that may cause QTc prolongation or induce Torsades de Pointes (See Appendix C, Table 1). Drugs listed in Appendix C, Table 2, that in the investigator s opinion cannot be discontinued are allowed; however, must be monitored closely with additional ECGs and laboratory assessments of electrolytes to ensure the patient s safety.
* Previous history of QTc prolongation with other medication.
* Congenital long QT syndrome
* QTc with Bazett's correction that is unmeasurable, or greater than or equal to 460 msec on screening ECG. If a patient has QTc greater than or equal to 460 msec on screening ECG, a second screen ECG may be repeated at least 24 hours apart. The average QTc from the 2 screening ECGs must be less than 460 msec in order for the patient to be eligible for the study. If the patient meets eligibility requiremen...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-12-29; Primary Completion 2014-02-27 (Actual); Study Completion 2014-02-27 (Actual)

PRIMARY OUTCOMES:
To establish the maximally tolerated dose of ZD6474 in patients with recurrent high-grade gliomas taking EIAED.

SECONDARY OUTCOMES:
To obtain preliminary information regarding the spectrum of toxicities, and to obtain pharmacokinetic data on ZD6474 administered to patients with recurrent high-grade gliomas taking EIAED.

CONTACTS AND LOCATIONS:
Overall Officials: Teri N Kreisl, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barker D, Wright E, Nguyen K, Cannon L, Fain P, Goldgar D, Bishop DT, Carey J, Baty B, Kivlin J, et al. Gene for von Recklinghausen neurofibromatosis is in the pericentromeric region of chromosome 17. Science. 1987 May 29;236(4805):1100-2. doi: 10.1126/science.3107130.
- [Background] Bigner SH, Bjerkvig R, Laerum OD. DNA content and chromosomal composition of malignant human gliomas. Neurol Clin. 1985 Nov;3(4):769-84. PMID 3001489
- [Background] Moss AR. Occupational exposure and brain tumors. J Toxicol Environ Health. 1985;16(5):703-11. doi: 10.1080/15287398509530780. PMID 4093991